CLINICAL TRIAL: NCT00557999
Title: Evaluation of the Effects of the Use of Mechanical Ventilation Weaning Protocol in the Coronary Care Unit: A Randomized Study
Brief Title: Mechanical Ventilation Weaning Protocol in the Coronary Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Base (Other)
Collaborators: Sao Jose do Rio Preto Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE-0009.0.140.000-06; C71050P
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Mechanical Ventilation; Cardiomyopathy
Keywords: Cardiology; Mechanical ventilation; Intensive care
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Other): Application of a weaning mechanical ventilation protocol
  Interventions: Other: Application of mechanical ventilation weaning protocol
- Control group (No Intervention)
  Interventions: Other: Application of mechanical ventilation weaning protocol

INTERVENTIONS:
Other: Application of mechanical ventilation weaning protocol — Application protocol for 8 months in experimental group

SUMMARY:
The following objectives were used for comparison: 1) primary objective: reintubation rate during hospitalization; 2) secondary objectives: length of hospitalization at the Coronary Care Unit; time from intubation to start of weaning; time from start of weaning to extubation; time from SBT and extubation; presence of respiratory infection in patients requiring reintubation; mortality of patients requiring reintubation.

DETAILED DESCRIPTION:
Once the cause leading to the need of MV was resolved, patients from both groups underwent a daily clinical evaluation in the mornings, to determine whether they were ready for mechanical ventilation weaning, according to the following clinical SBT criteria: 1) Cause of MV: resolution of the cause and abnormalities leading to MV; 2) neurological stability: patient awake, without or with minimal infusion of sedatives/narcotics, with effective cough and Glasgow scale ≥ 9; 3) cardiovascular stability: mean blood pressure (MBP) ≥ 60 mm Hg, without vasopressors or with low vasopressor doses, heart rate (HR) ≤ 140 / min, hemoglobin (Hb) ≥ 8,0 - 10,0 g/L, partial arterial oxygen pressure (PaO2) ≥ 60 mm Hg with fraction of inhaled oxygen (FiO2) ≤ 0.4, oxygenation index (PaO2 / FiO2) ≥ 150 - 300 without significant respiratory acidosis; 4) metabolic stability: temperature < 37.8° C (armpit) and lack of hydroelectrolytic disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized at the CCU with MV for over 24 hours;
* age over 18 years;
* both genders;
* patients capable of spontaneous ventilation;
* patients with indication for MV weaning.

Exclusion Criteria:

* conditions and/or circumstances that might result in difficulty to understand the informed consent (psychiatric disorder, alcohol or drug addiction, mental disability);
* patient denies to sign the informed consent;
* end-stage diseases and
* dependence on mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Measure: reintubation rates after mechanical ventilation weaning protocol | 48 hours after extubation

SECONDARY OUTCOMES:
Duration of mechanical ventilation weaning | within the first 7 days after indication of mechanical ventilation weaning

CONTACTS AND LOCATIONS:
Overall Officials: Lilia N Maia, phD, Study Director — Sao Jose do Rio Preto Medical School